CLINICAL TRIAL: NCT00974961
Title: Comparison of the Effects of Levobupivacaine and Bupivacaine on Heart Rate Variability in Spinal Anesthesia
Brief Title: Levobupivacaine on Heart Rate Variability (HRV) in Spinal Anesthesia
Acronym: HRV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shihyu,Chen / Attending Stuff, Attending Stuff of Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200903050M
Record Dates: First submitted 2009-09-07; First posted 2009-09-11 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Spinal Anesthesia
Keywords: Levobupivacaine; HRV; Spinal Anesthesia; Responses of ANS to these two drugs
MeSH Terms: interventions — Bupivacaine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levobupivacaine (Active Comparator): Lumbar puncture with Levobupivacaine for spinal anesthesia
  Interventions: Drug: bupivacaine, levobupivacaine
- Bupivacaine (Active Comparator): Lumbar puncture with Bupivacaine for spinal anesthesia
  Interventions: Drug: bupivacaine, levobupivacaine

INTERVENTIONS:
Drug: bupivacaine, levobupivacaine — intrathecal injection 15~20mg(for Levobupivacaine) or 10~15mg(for Bupivacaine) once

SUMMARY:
The purpose of this study is to compare if the effect of levobupivacaine on autonomic nervous system smaller than that of bupivacaine.

DETAILED DESCRIPTION:
Obtain the heart rate variability (in means and standard deviation, including the high frequency, low frequency and its ratio) data of before and after spinal anesthesia with ECG (and Heart Rate Variability Analyzer) in 2 groups. Meanwhile, record the blood pressure on each subject.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for spinal anesthesia

Exclusion Criteria:

* Allergic reaction to local anesthetics
* Coagulopathy
* Severe spinal deformity
* Cardiac diseases
* Metabolic diseases (such as DM, thyroid or adrenal diseases)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-12 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
HRV values | 5 minutes after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yu Chen, Study Chair
Locations (1):
- Department of Anesthesiology, National Taiwan University Hospital, Yun-Lin Branch, Yun-Lin County, Taiwan